CLINICAL TRIAL: NCT02403349
Title: Comparison of Peripheral and Cerebral Arterial Flow in Acute Ischemic Stroke: Fimasartan vs. Valsartan vs. Atenolol
Acronym: FAVOR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ajou University School of Medicine (Other)
Collaborators: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Ji Man Hong, Associate Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AJIRB-MED-CT4-12-049-HJM
Record Dates: First submitted 2015-03-12; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Blood Pressure; Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — fimasartan; Valsartan; Atenolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fimasartan (Experimental): fimasartan potassium 60mg, 1 tablet by mouth, every day Angiotensin ll receptor blocker
  Interventions: Drug: Fimasartan
- Valsartan (Active Comparator): valsartan 80mg, 1 tablet by mouth, every day angiotensin II receptor antagonists
  Interventions: Drug: Valsartan
- Atenolol (Active Comparator): atenolol 50mg, 1 tablet by mouth, every day beta-blocker
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Fimasartan
  Other Names: kanarb
  Arms: Fimasartan
Drug: Valsartan
  Other Names: Diovan
  Arms: Valsartan
Drug: Atenolol
  Other Names: tenormin
  Arms: Atenolol

SUMMARY:
Confirm central blood pressure reduction effect of Fimasartan, Valsartan and Atenolol and compare correlation with the measured peripheral (central blood pressure, pulse wave velocity, and flow-mediated dilation) and cerebral blood flow factors (transcranial doppler findings, cerebral blood flow volume) in acute ischemic stroke patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 30 years old
* Acute ischemic stroke patient who has corresponding DWI(diffusion- weighted imaging) lesion correlated with symptom
* after 7days, but within 28days from stroke onset
* Diagnosed with Hypertension
* hypertensive patients who taking anti-hypertensive drugs or SBP≥140mmHg
* Informed consent

Exclusion Criteria:

* Patients with hemorrhagic Stroke
* Patients with severe Stroke - over NIHss(National Institutes of Health stroke scale) 16
* Uncontrolled hypertension (SBP ≥200mmHg)
* Patients with history of allergic reaction to any angiotensin II antagonist
* Liver disease(more than double to normal level, SGOT(serum glutamic-oxaloacetic transaminase ), SGPT(serum glutamic-pyruvic transaminase ), total bilirubin)
* Renal disease(serum creatinine ≥2.0mg/dl)
* Anemia(Hb < 8mg/dl)
* Thrombocytopenia( < 10^3/ml)
* Patients with secondary hypertension
* Childbearing and breast-feeding women
* Otherwise inappropriate patients depending on the investigator's decision

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Central Blood pressure control | 12 weeks

SECONDARY OUTCOMES:
Blood pressure at the brachial artery | 12 weeks
Brachial-ankle pulse wave velocity (ba-PWV) | 12 weeks
  Ba-PWV is measured using ABI/PWV (VP-2000; Colin). This device has four cuffs that can be used to simultaneously measure blood pressure in both arms and both legs, and automatically calculate the ABI. It also records pulse waves with the sensors in the cuffs, computes the difference between transmission time in the arm and transmission time in the ankle, calculates the transmission distance from the right arm to each ankle according to body height, and thus computes the ba-PWV values from the transmission time and transmission distance.
Flow-mediated dilation (FMD) | 12 weeks
  FMD is measured as the brachial artery diameters at baseline and at maximum dilation after forearm ischemia for 5 minutes. FMD is calculated as the percentage of postischemic dilation.
Pulsatile index (PI) | 12 weeks
  We analyze the change of PIs in the middle cerebral artery at baseline and 90 Days on transcranial Doppler (TCD) Study in the same patient. The PI is automatically calculated on the TCD machine (PMD 150, Sphencer technologies, USA).
Cerebral blood flow (CBF) volume | 12 weeks
  CBF volume is measured by color-coded duplex sonography measuring total flow volumes of the internal carotid artery (ICAs) and vertebral artery (VAs).
Adverse Events | 12 weeks

REFERENCES:
- [Result] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. National Heart, Lung, and Blood Institute; National High Blood Pressure Education Program Coordinating Committee. Seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Hypertension. 2003 Dec;42(6):1206-52. doi: 10.1161/01.HYP.0000107251.49515.c2. Epub 2003 Dec 1. PMID 14656957
- [Result] Lewington S, Clarke R, Qizilbash N, Peto R, Collins R; Prospective Studies Collaboration. Age-specific relevance of usual blood pressure to vascular mortality: a meta-analysis of individual data for one million adults in 61 prospective studies. Lancet. 2002 Dec 14;360(9349):1903-13. doi: 10.1016/s0140-6736(02)11911-8. PMID 12493255
- [Result] Wiysonge CS, Bradley H, Mayosi BM, Maroney R, Mbewu A, Opie LH, Volmink J. Beta-blockers for hypertension. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD002003. doi: 10.1002/14651858.CD002003.pub2. PMID 17253471
- [Result] Heart Outcomes Prevention Evaluation Study Investigators; Yusuf S, Sleight P, Pogue J, Bosch J, Davies R, Dagenais G. Effects of an angiotensin-converting-enzyme inhibitor, ramipril, on cardiovascular events in high-risk patients. N Engl J Med. 2000 Jan 20;342(3):145-53. doi: 10.1056/NEJM200001203420301. PMID 10639539
- [Result] Lindholm LH, Ibsen H, Dahlof B, Devereux RB, Beevers G, de Faire U, Fyhrquist F, Julius S, Kjeldsen SE, Kristiansson K, Lederballe-Pedersen O, Nieminen MS, Omvik P, Oparil S, Wedel H, Aurup P, Edelman J, Snapinn S; LIFE Study Group. Cardiovascular morbidity and mortality in patients with diabetes in the Losartan Intervention For Endpoint reduction in hypertension study (LIFE): a randomised trial against atenolol. Lancet. 2002 Mar 23;359(9311):1004-10. doi: 10.1016/S0140-6736(02)08090-X. PMID 11937179
- [Result] Diener HC, Sacco R, Yusuf S; Steering Committee; PRoFESS Study Group. Rationale, design and baseline data of a randomized, double-blind, controlled trial comparing two antithrombotic regimens (a fixed-dose combination of extended-release dipyridamole plus ASA with clopidogrel) and telmisartan versus placebo in patients with strokes: the Prevention Regimen for Effectively Avoiding Second Strokes Trial (PRoFESS). Cerebrovasc Dis. 2007;23(5-6):368-80. doi: 10.1159/000100105. Epub 2007 Feb 26. PMID 17337887
- [Result] Schrader J, Luders S, Kulschewski A, Hammersen F, Plate K, Berger J, Zidek W, Dominiak P, Diener HC; MOSES Study Group. Morbidity and Mortality After Stroke, Eprosartan Compared with Nitrendipine for Secondary Prevention: principal results of a prospective randomized controlled study (MOSES). Stroke. 2005 Jun;36(6):1218-26. doi: 10.1161/01.STR.0000166048.35740.a9. Epub 2005 May 5. PMID 15879332
- [Result] Geeganage C, Tracy M, England T, Sare G, Moulin T, Woimant F, Christensen H, De Deyn PP, Leys D, O'Neill D, Ringelstein EB, Bath PM; for TAIST Investigators. Relationship between baseline blood pressure parameters (including mean pressure, pulse pressure, and variability) and early outcome after stroke: data from the Tinzaparin in Acute Ischaemic Stroke Trial (TAIST). Stroke. 2011 Feb;42(2):491-3. doi: 10.1161/STROKEAHA.110.596163. Epub 2010 Dec 23. PMID 21183747
- [Result] Oliveira-Filho J, Silva SC, Trabuco CC, Pedreira BB, Sousa EU, Bacellar A. Detrimental effect of blood pressure reduction in the first 24 hours of acute stroke onset. Neurology. 2003 Oct 28;61(8):1047-51. doi: 10.1212/01.wnl.0000092498.75010.57. PMID 14581662
- [Result] Sandset EC, Bath PM, Boysen G, Jatuzis D, Korv J, Luders S, Murray GD, Richter PS, Roine RO, Terent A, Thijs V, Berge E; SCAST Study Group. The angiotensin-receptor blocker candesartan for treatment of acute stroke (SCAST): a randomised, placebo-controlled, double-blind trial. Lancet. 2011 Feb 26;377(9767):741-50. doi: 10.1016/S0140-6736(11)60104-9. PMID 21316752
- [Result] Steckelings UM, Rompe F, Kaschina E, Unger T. The evolving story of the RAAS in hypertension, diabetes and CV disease: moving from macrovascular to microvascular targets. Fundam Clin Pharmacol. 2009 Dec;23(6):693-703. doi: 10.1111/j.1472-8206.2009.00780.x. Epub 2009 Oct 9. PMID 19817870
- [Result] Dzau VJ, Antman EM, Black HR, Hayes DL, Manson JE, Plutzky J, Popma JJ, Stevenson W. The cardiovascular disease continuum validated: clinical evidence of improved patient outcomes: part I: Pathophysiology and clinical trial evidence (risk factors through stable coronary artery disease). Circulation. 2006 Dec 19;114(25):2850-70. doi: 10.1161/CIRCULATIONAHA.106.655688. No abstract available. PMID 17179034
- [Result] NAVIGATOR Study Group; McMurray JJ, Holman RR, Haffner SM, Bethel MA, Holzhauer B, Hua TA, Belenkov Y, Boolell M, Buse JB, Buckley BM, Chacra AR, Chiang FT, Charbonnel B, Chow CC, Davies MJ, Deedwania P, Diem P, Einhorn D, Fonseca V, Fulcher GR, Gaciong Z, Gaztambide S, Giles T, Horton E, Ilkova H, Jenssen T, Kahn SE, Krum H, Laakso M, Leiter LA, Levitt NS, Mareev V, Martinez F, Masson C, Mazzone T, Meaney E, Nesto R, Pan C, Prager R, Raptis SA, Rutten GE, Sandstroem H, Schaper F, Scheen A, Schmitz O, Sinay I, Soska V, Stender S, Tamas G, Tognoni G, Tuomilehto J, Villamil AS, Vozar J, Califf RM. Effect of valsartan on the incidence of diabetes and cardiovascular events. N Engl J Med. 2010 Apr 22;362(16):1477-90. doi: 10.1056/NEJMoa1001121. Epub 2010 Mar 14. PMID 20228403
- [Result] Jankowski P, Kawecka-Jaszcz K, Czarnecka D, Brzozowska-Kiszka M, Styczkiewicz K, Loster M, Kloch-Badelek M, Wilinski J, Curylo AM, Dudek D; Aortic Blood Pressure and Survival Study Group. Pulsatile but not steady component of blood pressure predicts cardiovascular events in coronary patients. Hypertension. 2008 Apr;51(4):848-55. doi: 10.1161/HYPERTENSIONAHA.107.101725. Epub 2008 Feb 11. PMID 18268136
- [Result] Roman MJ, Devereux RB, Kizer JR, Lee ET, Galloway JM, Ali T, Umans JG, Howard BV. Central pressure more strongly relates to vascular disease and outcome than does brachial pressure: the Strong Heart Study. Hypertension. 2007 Jul;50(1):197-203. doi: 10.1161/HYPERTENSIONAHA.107.089078. Epub 2007 May 7. PMID 17485598
- [Result] Safar ME, Blacher J, Pannier B, Guerin AP, Marchais SJ, Guyonvarc'h PM, London GM. Central pulse pressure and mortality in end-stage renal disease. Hypertension. 2002 Mar 1;39(3):735-8. doi: 10.1161/hy0202.098325. PMID 11897754
- [Result] Roman MJ, Devereux RB, Kizer JR, Okin PM, Lee ET, Wang W, Umans JG, Calhoun D, Howard BV. High central pulse pressure is independently associated with adverse cardiovascular outcome the strong heart study. J Am Coll Cardiol. 2009 Oct 27;54(18):1730-4. doi: 10.1016/j.jacc.2009.05.070. PMID 19850215
- [Result] Williams B, Lacy PS, Thom SM, Cruickshank K, Stanton A, Collier D, Hughes AD, Thurston H, O'Rourke M; CAFE Investigators; Anglo-Scandinavian Cardiac Outcomes Trial Investigators; CAFE Steering Committee and Writing Committee. Differential impact of blood pressure-lowering drugs on central aortic pressure and clinical outcomes: principal results of the Conduit Artery Function Evaluation (CAFE) study. Circulation. 2006 Mar 7;113(9):1213-25. doi: 10.1161/CIRCULATIONAHA.105.595496. Epub 2006 Feb 13. PMID 16476843
- [Result] Dhakam Z, McEniery CM, Yasmin, Cockcroft JR, Brown MJ, Wilkinson IB. Atenolol and eprosartan: differential effects on central blood pressure and aortic pulse wave velocity. Am J Hypertens. 2006 Feb;19(2):214-9. doi: 10.1016/j.amjhyper.2005.08.007. PMID 16448896
- [Result] Neutel J, Weber M, Pool J, Smith D, Fitzsimmons S, Chiang YT, Gatlin M. Valsartan, a new angiotensin II antagonist: antihypertensive effects over 24 hours. Clin Ther. 1997 May-Jun;19(3):447-58; discussion 367-8. doi: 10.1016/s0149-2918(97)80129-4. PMID 9220209
- [Result] Takazawa K, Kobayashi H, Shindo N, Tanaka N, Yamashina A. Relationship between radial and central arterial pulse wave and evaluation of central aortic pressure using the radial arterial pulse wave. Hypertens Res. 2007 Mar;30(3):219-28. doi: 10.1291/hypres.30.219. PMID 17510503
- [Result] Yamashina A, Tomiyama H, Takeda K, Tsuda H, Arai T, Hirose K, Koji Y, Hori S, Yamamoto Y. Validity, reproducibility, and clinical significance of noninvasive brachial-ankle pulse wave velocity measurement. Hypertens Res. 2002 May;25(3):359-64. doi: 10.1291/hypres.25.359. PMID 12135313
- [Result] Lim MH, Cho YI, Jeong SK. Homocysteine and pulsatility index of cerebral arteries. Stroke. 2009 Oct;40(10):3216-20. doi: 10.1161/STROKEAHA.109.558403. Epub 2009 Jul 23. PMID 19628800
- [Result] Kim DH, Choi JH, Moon JS, Kim HJ, Cha JK. Association between the severity of cerebral small vessel disease, pulsatility of cerebral arteries, and brachial ankle pulse wave velocity in patients with lacunar infarction. Eur Neurol. 2010;64(4):247-52. doi: 10.1159/000319923. Epub 2010 Sep 11. PMID 20838053
- [Result] Hong JM, Lee JS, Shin DH, Yong SW. Hemodynamic impact of fetal-variant Willisian circle on cerebral circulation: a duplex ultrasonography study. Eur Neurol. 2011;65(6):340-5. doi: 10.1159/000327213. Epub 2011 May 19. PMID 21597296